CLINICAL TRIAL: NCT03312634
Title: A Phase 3, Efficacy and Safety Study of Oral Palovarotene for the Treatment of Fibrodysplasia Ossificans Progressiva (FOP)
Brief Title: An Efficacy and Safety Study of Palovarotene for the Treatment of Fibrodysplasia Ossificans Progressiva.
Acronym: MOVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clementia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVO-1A-301; 2017-002541-29 (EudraCT Number)
Record Dates: First submitted 2017-10-09; First posted 2017-10-18 (Actual); Results first posted 2023-03-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Fibrodysplasia Ossificans Progressiva
Keywords: Interventional study; Clinical trial phase 3; Efficacy and safety; Heterotopic ossification; Flare-up; Palovarotene; Retinoic acid receptor agonist; Retinoic acid receptor gamma agonist; Clementia; Myositis Ossificans Progressiva; Munchmeyer's Disease; FOP; FOP variants
MeSH Terms: conditions — Myositis Ossificans; Ossification, Heterotopic | interventions — Palovarotene

STUDY DESIGN:
Intervention Model Description: A multicenter, open-label study. NHS data (study PVO-1A-001) will be used as an external control in the analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Palovarotene Chronic/Flare-Up Regimen (Experimental): Participants received 5 mg palovarotene once daily for up to 48 months; and 20 mg palovarotene once daily for 28 days, followed by 10 mg for 56 days for flareups. (Dosing was adjusted for weight in skeletally immature subjects.)
  Interventions: Drug: Palovarotene

INTERVENTIONS:
Drug: Palovarotene — Palovarotene was taken orally once daily at approximately the same time each day following a meal.

SUMMARY:
Fibrodysplasia Ossificans Progressiva (FOP) is a rare, severely disabling disease characterized by heterotopic ossification (HO) often associated with painful, recurrent episodes of soft tissue swelling (flare-ups) that lead to ankyloses of major joints with cumulative and irreversible loss of movement and disability.

DETAILED DESCRIPTION:
One of the primary objectives was to evaluate the efficacy of palovarotene in decreasing new HO in participants with FOP as assessed by low-dose, whole body computed tomography (WBCT), excluding head, compared to untreated participants from Clementia's FOP natural history study (Study PVO-1A-001, NHS). The other primary objective was to evaluate the safety of palovarotene in participants with FOP.

This study was conducted in three parts. Part A was the main part of the study, Part B, the 2-year (24-month) extension and Part C was an up-to-2-year post last dose of study treatment follow-up for skeletally immature participants.

Participants in Part A and B received a chronic/flare-up dosing regimen of palovarotene for up to 4 years (48 months) as follows:

* Chronic treatment: orally administered 5 mg palovarotene once daily.
* Flare-up treatment: orally administered 20 mg palovarotene once daily for 4 weeks (28 days) followed by orally administered 10 mg palovarotene once daily for 8 weeks (56 days). Flare-up treatment may be extended until the Investigator determines that the flare-up has resolved.

Note that all dosing was weight-adjusted in skeletally immature participants (those under the age of 18 years with less than 90% skeletal maturity on hand/wrist x-rays performed at Screening).

In part C, participants who were enrolled in Parts A or B who discontinued the study and were skeletally immature were invited back to participate in the off-treatment safety follow-up. No new participants were enrolled into Part C.

ELIGIBILITY:
Key Inclusion Criteria:

* Written, signed, and dated informed subject/parent consent; and for subjects who are minors, age-appropriate assent (performed according to local regulations).
* Males or females at least 4 years of age.
* No flare-up symptoms within the past 4 weeks, including at the time of enrollment.
* Abstinent or using two highly effective forms of birth control.
* Accessible for treatment and follow-up; able to undergo all study procedures including low-dose WBCT (excluding head) without sedation.

Key Exclusion Criteria:

* Weight <10 kg.
* Concomitant medications that are strong inhibitors or inducers of cytochrome P450 (CYP450) 3A4 activity; or kinase inhibitors such as imatinib.
* Amylase or lipase >2x above the upper limit of normal (ULN) or with a history of chronic pancreatitis.
* Elevated aspartate aminotransferase or alanine aminotransferase >2.5x ULN.
* Fasting triglycerides >400 mg/dL with or without therapy.
* Female subjects who are breastfeeding.
* Subjects with uncontrolled cardiovascular, hepatic, pulmonary, gastrointestinal, endocrine, metabolic, ophthalmologic, immunologic, psychiatric, or other significant disease.
* Simultaneous participation in another clinical research study (other than palovarotene studies) within 4 weeks prior to Screening; or within five half-lives of the investigational agent, whichever is longer.
* Any reason that, in the opinion of the Investigator, would lead to the inability of the subject and/or family to comply with the protocol.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2022-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (16):
- United States (4):
  - University of California San Francisco, Division of Endocrinology and Metabolism, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Internal Medicine, Philadelphia, Pennsylvania
- Hospital Italiano de Buenos Aires, Tte General Juan Domingo Peron 4190, Buenos Aires, Argentina
- Australia (2):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Queensland University of Technology, Woolloongabba, Queensland
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil
- Canada (2):
  - Hospital for Sick Children, 555 University Avenue, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Groupe Hospitalier Necker Enfants Malades, Paris, France
- Istituto Giannina Gaslini, Genoa, Liguria, Italy
- The University of Tokyo Hospital, Tokyo, Bunkyo-ku, Japan
- Hospital Universitari i Politècnic La Fe, Unidad de Reumatología Pediatrica, Valencia, Avinguda de Fernando Abril Martorell, Nº 106, Spain
- Norrlands Universitetssjukhus, Umeå, Sweden
- Royal National Orthopaedic Hospital, Brockely Hill, Stanmore, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shimono K, Tung WE, Macolino C, Chi AH, Didizian JH, Mundy C, Chandraratna RA, Mishina Y, Enomoto-Iwamoto M, Pacifici M, Iwamoto M. Potent inhibition of heterotopic ossification by nuclear retinoic acid receptor-gamma agonists. Nat Med. 2011 Apr;17(4):454-60. doi: 10.1038/nm.2334. Epub 2011 Apr 3. PMID 21460849
- [Derived] Lindborg CM, Al Mukaddam M, Baujat G, Cho TJ, De Cunto CL, Delai PLR, Eekhoff EMW, Haga N, Hsiao EC, Morhart R, de Ruiter R, Scott C, Seemann P, Szczepanek M, Tabarkiewicz J, Pignolo RJ, Kaplan FS. Most Fractures Treated Nonoperatively in Individuals With Fibrodysplasia Ossificans Progressiva Heal With a Paucity of Flareups, Heterotopic Ossification, and Loss of Mobility. Clin Orthop Relat Res. 2023 Dec 1;481(12):2447-2458. doi: 10.1097/CORR.0000000000002672. Epub 2023 May 8. PMID 37156007
- [Derived] Pignolo RJ, Hsiao EC, Al Mukaddam M, Baujat G, Berglund SK, Brown MA, Cheung AM, De Cunto C, Delai P, Haga N, Kannu P, Keen R, Le Quan Sang KH, Mancilla EE, Marino R, Strahs A, Kaplan FS. Reduction of New Heterotopic Ossification (HO) in the Open-Label, Phase 3 MOVE Trial of Palovarotene for Fibrodysplasia Ossificans Progressiva (FOP). J Bone Miner Res. 2023 Mar;38(3):381-394. doi: 10.1002/jbmr.4762. Epub 2023 Jan 25. PMID 36583535
- See also: Website for the International FOP Association — http://ifopa.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3, open-label study conducted in adult and pediatric participants with fibrodysplasia ossificans progressiva (FOP) at 16 centers in 11 countries (Argentina, Australia, Brazil, Canada, France, Italy, Japan, Spain, Sweden, the United Kingdom, and the US) between 30 November 2017 and 07 September 2022.
Pre-assignment Details: This study included 3 parts: Part A, the main part of the study, Part B, the 24-month extension and Part C, up to 2 year post last dose of study treatment follow-up. A total of 107 participants were enrolled and treated in this study. Data from participants in PVO-1A-001 were used as an external control for only primary endpoint of this study. Hence, data for participants in PVO-1A-001 are reported in participant flow, baseline characteristics and adverse events section only.
Groups:
- Palovarotene: Participants were administered 5 milligram (mg) palovarotene orally once daily up to 48 months. Participants with flare-up symptoms or traumatic events received palovarotene 20 mg once daily for 4 weeks after the flare-up confirmation by the Investigator. Followed by palovarotene 10 mg once daily for 8 weeks.
- Untreated (PVO-1A-001): Participants from study PVO-1A-001 (NCT02322255) were included with FOP caused by the R206H mutation and with baseline data. Participants were not administered palovarotene in this study and only compared as external control.
Period: Overall Study
Arm/Group | Palovarotene | Untreated (PVO-1A-001)
Started | 107 | 114
Completed | 49 | 33
Not Completed | 58 | 81
Not completed — Adverse Event | 11 | 0
Not completed — Sponsor request | 2 | 0
Not completed — Withdrawal by Subject | 31 | 9
Not completed — Enrolled in an interventional study | 0 | 52
Not completed — Enrolled in an interventional study at time of a flare-up | 0 | 9
Not completed — Death | 0 | 1
Not completed — Non-compliance | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Enrolled into non-interventional study | 0 | 5
Not completed — Worsening clinical condition | 0 | 1
Not completed — Participant did not want to travel | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Other | 13 | 0

BASELINE CHARACTERISTICS:
Population: The Principal Safety Set (Principal SS) included all enrolled participants in the Principal Enrolled Population (Principal EP) set [ie, participants with the R206H activin receptor type IA (ACVR1) mutation] receiving at least 1 dose of palovarotene in study PVO-1A-301. The Full Analysis Set (FAS) included all participants in the Enrolled Analysis Set with FOP caused by the R206H mutation and who had baseline data in study PVO-1A-001 (NCT02322255).
Groups:
- Palovarotene: Participants were administered 5 mg palovarotene orally once daily up to 48 months. Participants with flare-up symptoms or traumatic events received palovarotene 20 mg once daily for 4 weeks after the flare-up confirmation by the Investigator. Followed by palovarotene 10 mg once daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Palovarotene | Untreated (PVO-1A-001) | Total
Number analyzed (Participants) | 99 | 114 | 213
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 75 | 70 | 145
  Between 18 and 65 years | 24 | 44 | 68
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 52 | 98
  Male | 53 | 62 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 23 | 42
  Not Hispanic or Latino | 69 | 73 | 142
  Unknown or Not Reported | 11 | 18 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 70 | 84 | 154
  Black or African American | 1 | 0 | 1
  Asian | 9 | 8 | 17
  American Indian or Alaska Native | 0 | 1 | 1
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Multiple | 6 | 2 | 8
  Other | 1 | 4 | 5
  Unknown | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Annualized New Heterotopic Ossification (HO)
Description: The annualized new HO was assessed by low-dose, whole body computed tomography (WBCT), excluding head. The weighted linear mixed effect method without square-root transformation and negatives included was used for annualized new HO analysis.
Time Frame: Baseline (within one month of screening/Day 1) and up to 24 months
Population: The Principal FAS includes all enrolled participants in the Principal EP who had a baseline HO volume measurement and at least 1 post-baseline HO volume measurement in study PVO-1A-301. For study PVO-1A-001, the Principal FAS included participants enrolled in study PVO-1A-001 with available baseline and at least 1 post-baseline HO volume measurement. Study PVO-1A-001 was used as an external control.
Measure: Mean (Standard Error); unit: cubic millimeters (mm^3)
Arm/Group | Palovarotene | Untreated (PVO-1A-001)
Number analyzed (Participants) | 97 | 101
cubic millimeters (mm^3) | 9427.1 (3084.0) | 23720.2 (4850.0)

2. Secondary Outcome: Percentage of Participants With Any New HO
Description: The new HO was assessed by WBCT scan. The percentage of participants with any new HO (volume > 0 mm^3) were analyzed using the Bayesian distribution. Results are presented for overall ITT period.
Time Frame: From Baseline (Day 1) up to end of 4-year follow-up period (approximately 57 months)
Population: The Principal FAS included all enrolled participants in the Principal EP who had a baseline HO volume measurement and at least 1 post-baseline HO volume measurement in study PVO-1A-301.
Measure: Number; unit: percentage of participants
Arm/Group | Palovarotene
Number analyzed (Participants) | 97
percentage of participants | 83.5

3. Secondary Outcome: Number of Body Regions With New HO
Description: All participants were analyzed for number of body regions with any new HO (new HO > 0 mm^3). The presence of HO across various body regions was analyzed using WBCT scan. Results are presented for overall ITT period
Time Frame: From Baseline (Day 1) up to end of 4-year follow-up period (approximately 57 months)
Population: The Principal FAS included all enrolled participants in the Principal EP who had a baseline HO volume measurement and at least 1 post-baseline HO volume measurement in the study PVO-1A-301. Only data from the participants analyzed were reported.
Measure: Mean (Standard Deviation); unit: body regions
Arm/Group | Palovarotene
Number analyzed (Participants) | 81
body regions | 3.0 (1.68)

4. Secondary Outcome: Percentage of Participants With Flare-Ups
Description: Flare-up as an event with one or more flare-up symptoms, and regardless of flare-up symptom onset. Flare-up was evaluated remotely, or by telephone or video-conferencing, unless the Investigator deemed that a site visit was necessary.
Time Frame: Month 12
Population: The Principal SS included all enrolled participants in the Principal EP set (ie, participants with the R206H ACVR1 mutation) receiving at least 1 dose of palovarotene in study PVO-1A-301. Only data from the participants analyzed at Month 12 reported.
Measure: Number; unit: percentage of participants
Arm/Group | Palovarotene
Number analyzed (Participants) | 99
percentage of participants | 64.6

5. Secondary Outcome: Ratio of Flare-Up Per Participant-Month of Exposure
Description: Flare-up as an event with one or more flare-up symptoms, and regardless of flare-up symptom onset. Flare-up was evaluated remotely, or by telephone or video-conferencing, unless the Investigator deemed that a site visit was necessary. The flare-up rate per participant-month exposure was analyzed using a negative binomial regression. Results are presented for overall ITT period.
Time Frame: From Baseline (Day 1) up to end of 4-year follow-up period (approximately 57 months)
Population: The Safety analysis set included all enrolled participants who received at least 1 dose of palovarotene in study PVO-1A-301.
Measure: Mean (Standard Deviation); unit: ratio of flare-up
Arm/Group | Palovarotene
Number analyzed (Participants) | 107
ratio of flare-up | 0.2 (0.40)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are collected from first date of palovarotene intake up to end of 4-year follow-up period (approximately 57 months) for study PVO-1A-301. For study PVO-1A-001, adverse events (AEs) were collected from study day 1 up to approximately 37 months. While no pharmacological intervention was applied in this observational study (PVO-1A-001), safety issues resulting only from any study-related procedure were recorded as AEs. MedDRA version 21.0 for PVO-1A-001 study.
Description: The Safety analysis set included all enrolled participants who received at least 1 dose of palovarotene in study PVO-1A-301. The FAS included all participants in the Enrolled Analysis Set with FOP caused by the R206H mutation and who had baseline data in study PVO-1A-001.
Groups:
- Palovarotene 5 mg: Participants were administered 5 mg palovarotene orally once daily up to 48 months.
- Palovarotene 20/10 mg: Participants with flare-up symptoms or traumatic events received palovarotene 20 mg once daily for 4 weeks after the flare-up confirmation by the Investigator. Followed by palovarotene 10 mg once daily for 8 weeks.
- Untreated (PVO-1A-001): Participants from study PVO-1A-001 (NCT02322255) were included with FOP caused by the R206H mutation and with baseline data. Participants were not administered palovarotene in this study and only compared as external control. While no pharmacological intervention was applied in this observational study, safety issues resulting only from any study-related procedure were recorded as AEs.
Arm/Group | Palovarotene 5 mg | Palovarotene 20/10 mg | Untreated (PVO-1A-001)
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/81 | 1/114
Serious Adverse Events (participants affected / at risk) | 34/107 | 19/81 | 0/114
Other Adverse Events (participants affected / at risk) | 105/107 | 77/81 | 0/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palovarotene 5 mg (N=107) | Palovarotene 20/10 mg (N=81) | Untreated (PVO-1A-001) (N=114)
Epiphyses Premature Fusion (Musculoskeletal and connective tissue disorders) | 11 (11) | 10 (10) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Epiphyseal Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mycoplasma Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Condition Aggravated (General disorders) | 2 (2) | 3 (3) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Aneurysmal bone cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 10 (10) | 2 (2) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palovarotene 5 mg (N=107) | Palovarotene 20/10 mg (N=81) | Untreated (PVO-1A-001) (N=114)
Dry skin (Skin and subcutaneous tissue disorders) | 60 (95) | 37 (77) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (23) | 21 (28) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 15 (24) | 26 (40) | 0
Pruritus (Skin and subcutaneous tissue disorders) | 19 (29) | 14 (16) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 25 (40) | 11 (22) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 11 (15) | 16 (21) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 11 (14) | 11 (23) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 6 (9) | 5 (6) | 0 (0)
Rash generalized (Skin and subcutaneous tissue disorders) | 6 (9) | 4 (5) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (8) | 0 (0)
Lip Dry (Gastrointestinal disorders) | 37 (38) | 17 (17) | 0 (0)
Chapped Lips (Gastrointestinal disorders) | 6 (7) | 10 (11) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (14) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (9) | 3 (3) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 3 (3) | 8 (13) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 23 (30) | 6 (7) | 0 (0)
Nasopharyngitis (Infections and infestations) | 14 (26) | 9 (12) | 0 (0)
Paronychia (Infections and infestations) | 9 (13) | 10 (15) | 0 (0)
Ear Infection (Infections and infestations) | 5 (5) | 6 (7) | 0 (0)
Otitis Media (Infections and infestations) | 6 (7) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (8) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 6 (6) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 (49) | 15 (24) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 21 (33) | 9 (13) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (9) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (13) | 3 (4) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 5 (5) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 9 (12) | 6 (6) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 8 (11) | 9 (13) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 10 (12) | 7 (12) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (14) | 3 (3) | 0 (0)
Dry Eye (Eye disorders) | 8 (8) | 11 (14) | 0 (0)
Headache (Nervous system disorders) | 10 (13) | 7 (7) | 0 (0)
Seasonal Allergy (Immune system disorders) | 7 (8) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 6 (8) | 4 (5) | 0 (0)
Influenza (Infections and infestations) | 7 (7) | 4 (4) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 6 (9) | 3 (3) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 3 (3) | 6 (7) | 0 (0)
Bone density decreased (Investigations) | 8 (8) | 5 (5) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 5 (5) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 6 (7) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 16 (21) | 11 (19) | 0 (0)

LIMITATIONS AND CAVEATS:
A valid comparison of AEs from observational study (PVO-1A-001) was not made since AEs were only captured as related to study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT03312634/Prot_002.pdf
  • Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT03312634/SAP_003.pdf